CLINICAL TRIAL: NCT07005362
Title: Feasibility of Use of Fitbit, Brief DSMES, and Targeted Text Messaging in Sedentary Adults With Type 2 Diabetes in Primary Care Settings
Brief Title: Fitbit and AI Chatbot in Sedentary Primary Care Patients With T2D
Acronym: FIT T2D
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Academy of Family Physicians (Other)
Responsible Party: Sponsor
Other Study IDs: 24-2577
Record Dates: First submitted 2025-05-23; First posted 2025-06-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Mellitus (T2DM); T2DM (Type 2 Diabetes Mellitus); T2D; T2DM; Remote Patient Monitoring; Artificial Intelegence
Keywords: type 2 diabetes; artificial intelligence; fitbit; primary care; remote patient monitoring; physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: Fitbit and AI Chatbot: Participants will wear their Fitbit devices daily and receive personalized messages from the AI Chatbot weekly with setting a new exercise goal based on their previous week's activity level. Additionally, they can engage with the AI Chatbot through text message for further support, education, and goal setting. Participants will interact throughout the week on completing their goal or where they might improve.
  Interventions: Behavioral: Fitbit and AI Chatbot
- Active Comparator: Controls: The control group will be established through a rigorous retrospective chart review of patients with type 2 diabetes who meet the study's inclusion criteria but have not participated in the intervention.
  Interventions: Other: Routine Care

INTERVENTIONS:
Behavioral: Fitbit and AI Chatbot — Participants will wear their Fitbit devices daily for 12-weeks and will receive personalized messages from the AI Chatbot every week with a new exercise recommendation based on their previous week's activity level. Additionally, they can engage with the AI Chatbot through text message for further support and education.
  Groups: Experimental: Fitbit and AI Chatbot
Other: Routine Care — The control group will consist of patients with type 2 diabetes who meet the study's inclusion criteria but have not participated in the intervention.
  Groups: Active Comparator: Controls

SUMMARY:
The goal of this observational study is to evaluate the feasibility and acceptability of a 12-week intervention utilizing a Fitbit and artificial intelligence (AI)-delivered diabetes self-management education and support (DSMES) with tailored text messages.

The main question it aims to answer is:

Does providing a wearable fitness and activity tracker plus AI-tailored and DSMES improve clinical outcomes for patients with type 2 diabetes?

Participants will complete a baseline visit, wear a Fitbit and answer text messages for 12-weeks, and complete by a final visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes per investigator discretion
* No more than 20% of the sample will have A1c < 7.5% (confirmed by medical record review or an A1c completed within 3 months of the screening visit)
* Age ≥18 years and ≤ 80 years
* Does not meet ADA guidelines for physical activity (< 150 minutes of aerobic exercise per week defined as any activity where the participant can talk but not sing)
* Has a smartphone compatible with a Fitbit

Exclusion Criteria:

* Completing more than 60 minutes of moderate to vigorous activity per week defined as activity where you cannot sing (moderate) or can't say more than a few words without gasping for breath (vigorous)(14)
* Any medical condition which, in the opinion of the investigator, would put the participant at an unacceptable safety risk, such as untreated malignancy, unstable cardiac disease, unstable or end-stage renal disease, and/or eating disorders.
* Current or known history of coronary artery disease that is not stable with medical management, including unstable angina, or angina that prevents moderate exercise despite medical management, or a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass grafting within the previous 12- months
* Any planned surgery during the study which could be considered major in the opinion of the investigator
* Blood disorder or dyscrasia within 3 months before screening, or the use of hydroxyurea, which, in the investigator's opinion, could interfere with the determination of HbA1c
* Has taken oral or injectable steroids within the past 8 weeks or plans to take oral or injectable steroids during the study, as they may interfere with the determination of HbA1c.
* Planning to move from Colorado within 3 months
* Current Pregnancy or planning on pregnancy in the next 3 months
* Unable to safely comply with study procedures and reporting requirements (e.g. impairment of vision that impacts ability to see FitBit, impaired memory)
* Unable to speak English as this is a small feasibility study that does not have the resources to adapt the intervention for Spanish
* Current participation in another diabetes-related clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care adult patients diagnosed with type 2 diabetes who do not meet ADA guidelines for physical activity (< 150 minutes of aerobic exercise per week defined as any activity where the participant can talk but not sing).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | 6 months
  Recruitment of 36 adults within 6 months.
Feasibility - Retainment | 6 months
  Retainment of 85% of participants for post-assessments.
Feasibility - Fitbit wear | 12 Weeks
  Fitbit wear ≥ 5 days/week > 12 hours per day, wear at night > 3 nights/week.
Feasibility - Text message responses | 12 Weeks
  Responding to 80% of text messages when prompted.
Feasibility - Technical issues | 12 Weeks
  Participation with ≤10% technical issues (battery life, data sync between device and app/dashboard, device failure).
Acceptability - Participant Experience and Satisfaction | 12 Weeks
  Obtaining > 60% satisfaction from participants via a satisfaction survey.

SECONDARY OUTCOMES:
Change in HbA1c | 12 Weeks
  Change in HbA1c from baseline to post-intervention.
Change in Body Mass Index | 12 Weeks
  Change in Body Mass Index (BMI) from baseline to post-intervention.
Change in lipid panel | 12 Weeks
  Change in lipid panel from baseline to post-intervention.
Change in weight | 12 Weeks
  Change in weight from baseline to post-intervention.
Change in blood pressure | 12 Weeks
  Change in blood pressure from baseline to post-intervention.
Change in diabetes distress | 12 Weeks
  Change in diabetes distress as measured by the T2-DDAS: The Type 2 Diabetes Distress Assessment System from baseline to post-intervention.
Experience with technology | 12 Weeks
  Patient experience with technology as measured via the System Usability Scale (SUS).
Experience with technology | 12 Weeks
  Patient experience with technology as measured via the FACETS Comfort with Technology assessment.
Cost | Weekly, 12 weeks
  Cost of delivering remote patient monitoring intervention as measured via time-diaries and patient logs.
Revenue | Weekly, 12 weeks
  Revenue modeling from practice perspective of remote patient monitoring intervention as measured via staff and patient time logs.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Kramer, DO, MPH, Principal Investigator — University of Colorado Anschutz Medical School
Locations (1):
- University of Colorado, Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided